CLINICAL TRIAL: NCT01841294
Title: NK Activity Modulation by Intravenous Lidocaine During Laparoscopic Colorectal Surgery
Brief Title: NK Activity Modulation Induced by Intravenous Lidocaine During Colorectal Laparoscopic Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Louis-Philippe Fortier, Principal investigator, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 11077
Record Dates: First submitted 2013-02-27; First posted 2013-04-26 (Estimated); Last update posted 2013-04-26 (Estimated); Status verified 2012-01

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravenous Lidocaine (Experimental): Patients undergoing laparoscopic surgery for resection of colorectal cancer will benefit of an infusion of intravenous lidocaine from the induction of anesthesia untill one hour after PACU admission
  Interventions: Drug: Intravenous Lidocaine
- Placebo (Placebo Comparator): Infusion of normal saline form the induction of anaesthesia untill one hour after PACU admission
  Interventions: Drug: Normal saline infusion

INTERVENTIONS:
Drug: Intravenous Lidocaine — Lidocaine infusion: 1.5 mg/kg bolus on 10 minutes (maximum 150 mg) followed by 1.5 mg/kg/h
  Other Names: Chlorydrate de Lidocaine 2%
  Arms: Intravenous Lidocaine
Drug: Normal saline infusion — Normal saline infusion: 1.5 mg/kg bolus on 10 minutes (maximum 150 mg) followed by 1.5 mg/kg/h
  Arms: Placebo

SUMMARY:
Surgical resection is the best treatment option for colorectal cancer. Despite this radical approach, recurrences within five years are still common. Several authors have proposed that the immunosuppressive state surrounding the perioperative period was a key element of cancer cells spread.

A particular subtype of T lymphocytes, the Natural Killer cells (NKs), is the main actor of the innate immune system. Several factors of the perioperative period can reduce activity of NKs such as stress, pain, opioids and general anaesthetics.

Lidocaine is a local anaesthetic that has been widely used intravenously for abdominal surgeries. Intravenous lidocaine has been shown to reduce pain scores, morphine consumption, ileus time and length of stay in major colorectal surgeries. It reduced markers of systemic inflammation as well.

The authors hypothesize that the use of intravenous lidocaine during laparoscopic surgeries for colorectal cancer resection will preserve NKs activity.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for resection of colorectal cancer under laparoscopic surgery
* American Society of Anesthesiologists class I-III.
* The subject is able to understand the study objectives, the experimental protocol and procedures, and is capable of providing an informed consent.

Exclusion Criteria:

* Subjects allergic to any of the study drugs.
* BMI > 35 kg/m2.
* Severe renal or hepatic failure.
* Pregnancy.
* Emergent procedure.
* Heart failure NYHA > III.
* Systolic blood pressure < 90 mmHg.
* Advanced heart block (unless patient has a pacemaker).
* Unstable angina and/or myocardial infarction within past 6 weeks.
* FEV1 ≤ 0.8 L.
* Oxygen-dependent patient.
* Electrocardiographic abnormalities
* Treatment with immunosupressive drugs, corticosteroids, NSAIDS, antiarythmic
* Morphine intolerance or allergy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Dosage of NKs activity after surgery | compare the activity of NK cells on day 1 and day 3 after surgery
  Dosage of NKs activity after surgery

SECONDARY OUTCOMES:
Pain scores | pain scores from the PACU to the 3rd day after surgery
  From the PACU to the 3rd day after surgery
Morphine consumption | From the PACU to the 3rd day after surgery
  Morphine consumption from the PACU to the 3rd day after surgery
Ileus time | Day 1 and Day 3 after surgery
  time to get flattus after surgery
Surgical complications | Within 3 days after surgery
  Infections, leakage, abcess
Fentanyl dose | Operative time
  Cumulative dose of fentanyl needed for the surgery
Nausea and vomiting | From the PACU to the 3rd day after surgery
  Nausea and vomiting from the PACU to the 3rd day after surgery
Major adverses events | Start of the surgery untill one hour after PACU ad;ission
  Hypotension, heart rythm blocks, tachycarida, bradycardia

CONTACTS AND LOCATIONS:
Overall Officials: Louis-Philippe Fortier, M.D., Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Hôpital Maisonneuve Rosemont, Montreal, Quebec, Canada